CLINICAL TRIAL: NCT03413163
Title: Ultrasound Guided Erector Spinae Plane Block for Postoperative Analgesia in Retropubic Radical Prostatectomy Patients; Randomised, Controlled Prospective Study
Brief Title: Ultrasound Guided Bilateral Erector Spinae Plane Block in Retropubic Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Özgür Şentürk, M.D., assistant professor, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maltepe University
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Pain
Keywords: Ultrasound Guided Erector Spinae Plane Block; postoperative pain; retropubic radical prostatectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Sham Comparator): Peroperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed.
  Intervention: Other: Standard Pain Followup and Monitorization
  Interventions: Other: Standard Pain Followup and Monitorization
- ESP block (Experimental): In addition to routine analgesic protocol; before anaesthesia induction; bilateral ultrasound guided erector spinae plane block (ESP) (intervention) will be performed via USG guidance at Th9 level.Standard Pain Followup and Monitorization will be performed.
  Interventions:
  Procedure: Ultrasound guided erector spinae plane block Other: Standard Pain Followup and Monitorization
  Interventions: Drug: Ultrasound guided erector spinae plane block; Other: Standard Pain Followup and Monitorization

INTERVENTIONS:
Drug: Ultrasound guided erector spinae plane block — A high-frequency linear ultrasound transducer will be placed in a longitudinal parasagittal orientation 3 cm lateral to T9 spinous process. The erector spinae muscles will be identified superficial to the tip of T9 transverse process. The patient's skin will be anesthetized with 2% lidocaine. A 17-gauge 8-cm needle will be inserted using an in-plane superior-to-inferior approach to place the tip into the fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting erector spinae muscle off the bony shadow of the transverse process. A total of 30 mL of 0.375% bupivacaine will be injected (maximum of 3mg/kg).
  Arms: ESP block
Other: Standard Pain Followup and Monitorization — Numeric Rating Scale (NRS) pain score will be recorded from 20th minute in recovery room followed by 1.-3.-6.-12.-18.-24.hours. Intravenous meperidine administration at 0.5 mg / kg rescue analgesia was determined in patients with a NSR score of 6 and over in the postoperative collection room. It is planned that the patient will continue to follow the hourly NRS score in ward. Intramuscular diclofenac will be administered in this period if NRS 6 and if it is over, intravenous 0.5 mg / kg meperidine will be administered if NRS score is 6 or more after 2 hours. Salvage analgesic needs and times will be noted in detail, and the use of rescue analgesics, as well as NRS scores at designated hours, will be kept in a statistical evaluation.

SUMMARY:
This study will define the postoperative analgesic effect of ESP block via amount of patient-controlled analgesia (PCA) and postoperative analgesic consumption (such as routinely and rescue analgesics) and compare the control group patients with retropubic radical prostatectomy .

DETAILED DESCRIPTION:
Open retropubic prostatectomy is a surgical method that is applied in cases of benign prostatic hypertrophy and prostate cancer which is not suitable for surgical treatment with closed method. This method is commonly used among urological procedures which are open surgical procedures. Patients after this procedure often complain of excessive pain. Non-steroidal anti-inflammatory agents and opioids are used for postoperative analgesia. In addition, in the past decade, in the guideline of ultrasonography, peripheral block types have been described that demonstrate analgesic activity in open prostatectomies as well as many operations on the development of regional anesthesia and analgesia techniques. The ultrasonography guideline reported that the transverse abdominal plane (TAP) block provides effective analgesia in these cases. The ESP block is a new block for the treatment of thoracic neuropathic pain. In the following process; ESP block thoracic and breast surgery, bariatric surgery, and upper abdominal surgeons have also been reported to provide effective postoperative analgesia.

The standard practice for post-operative pain management for retropubic radical prostatectomy in Maltepe University Hospital consists of routine intravenous analgesic and rescue analgesics and in combination with patient-controlled analgesia (PCA).

The application of erector spinae plane (ESP) block technique under ultrasonography guideline under sedoanalgesia in patients who will undergo retropubic prostatectomy with open method should determine the effect on the patient's pain level in the first 24 hours after operation.

ELIGIBILITY:
Inclusion Criteria:

Elective retropubic radikal prostatectomy, ASA status 1-2

Exclusion Criteria:

* Patient refusal
* Contraindications to regional anesthesia
* Known allergy to local anesthetics
* Bleeding diathesis
* Use of any anti-coagulants
* Inability to provide informed consent
* Severe kidney or liver disease
* Inability to operate PCA system
* Patient with psychiatric disorders

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Changes in Numeric Rating Scale (NRS) | 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
analgesic consumption | 24 hours
  Tramadol consumption in Patient Controlled Analgesia device and additional and rescue analgesic using

CONTACTS AND LOCATIONS:
Overall Officials: ozgur senturk, ass prof, Study Chair — maltepe university faculty of medicine
Locations (1):
- Maltepe University Medical Faculty, Istanbul, Feyzullah No:39, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

REFERENCES:
- [Result] Restrepo-Garces CE, Chin KJ, Suarez P, Diaz A. Bilateral Continuous Erector Spinae Plane Block Contributes to Effective Postoperative Analgesia After Major Open Abdominal Surgery: A Case Report. A A Case Rep. 2017 Dec 1;9(11):319-321. doi: 10.1213/XAA.0000000000000605. PMID 28727597
- [Result] Elkassabany N, Ahmed M, Malkowicz SB, Heitjan DF, Isserman JA, Ochroch EA. Comparison between the analgesic efficacy of transversus abdominis plane (TAP) block and placebo in open retropubic radical prostatectomy: a prospective, randomized, double-blinded study. J Clin Anesth. 2013 Sep;25(6):459-65. doi: 10.1016/j.jclinane.2013.04.009. Epub 2013 Aug 17. PMID 23965191
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016